CLINICAL TRIAL: NCT02263521
Title: Physician Work Motivation: A Measure Validation Study
Brief Title: Understanding Physician Work Motivation
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: American Medical Association (Other)
Collaborators: American Medical Group Association (Other); Illinois Institute of Technology (Other); Advocate Physician Partners (Unknown); University of California, San Francisco (Other); University of Rochester (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Audiey Kao, MD, PhD, Vice President, Ethics, American Medical Association
Other Study IDs: AMAHSA0901
Record Dates: First submitted 2014-09-28; First posted 2014-10-13 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Physician Work Motivation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- physicians: Nationally-representative sample of physicians in all specialties who have direct or indirect patient care responsibilities
  Interventions: Other: No intervention employed. Study is based on a cross-sectional observational design.
- resident physicians: Nationally-representative of resident physicians in all specialties
  Interventions: Other: No intervention employed. Study is based on a cross-sectional observational design.
- medical students: Nationally-representative sample of 4th year medical students in all US allopathic medical schools.
  Interventions: Other: No intervention employed. Study is based on a cross-sectional observational design.

INTERVENTIONS:
Other: No intervention employed. Study is based on a cross-sectional observational design.

SUMMARY:
Development and validation of a measure of physician work motivation.

DETAILED DESCRIPTION:
Not that long ago, most physicians were solo practitioners. Today, more physicians are working in large, integrated delivery systems, and many are employed by hospitals and multispecialty group practices. These dramatic changes in the physician work environment raise important questions on how evolving physician payment and care delivery models support or undermine your motivation and ability to deliver high-quality patient care.

To evaluate the impact of workplace changes on what motivates physician to deliver good patient care, this study aims to develop an accurate measure of physician work motivation. Simultaneously, the investigators plan to test hypotheses on the role of various workplace and psychological factors in physicians' work motivation. Namely, the investigators hypothesize that:

20 to 25% of the variance in work motivation is explained by psychological needs satisfaction; 5 to 10% of the variance in self-reported overall health status and depression is explained by work motivation; 5% of the variation in work motivation is explained by work that is seen as a calling; and 5 to 10% of the variation in medicine viewed as a calling is explained by the learning environment.

ELIGIBILITY:
Inclusion Criteria:

* practicing physicians in all medical specialties
* resident physicians in all medical specialties
* fourth year medical students in US allopathic medical schools

Exclusion Criteria:

* physicians without an active medical license.
* resident physicians without an active medical license.
* fourth year medical students in US osteopathic medical schools

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population #1 includes practicing physicians in all medical specialties. Population #2 includes resident physicians in all medical specialties. Population #3 includes fourth year medical students in all US allopathic medical schools.
Sampling Method: Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-05 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Internalization of work motivation (self-reported) | Up to 4 months
  Composite measure comprised of 15 items using 7-point Likert-type response categories (not at all true-very true) to assess extent of psychological internalization of work motivation

SECONDARY OUTCOMES:
Psychological needs satisfaction at work (self-reported) | Up to 4 months
  Composite measure comprised of 12 statements using 7-point Likert-type response categories (not at all true-very true) to assess perceived fulfillment of needs for autonomy, self-efficacy/competence, relatedness, and purpose in work context
Overall health status (self-reported) | Up to 4 months
  Proportion of respondents reporting own overall health as "excellent," "very good," or "good" vs. "fair" or "poor"
Depression (self-reported) | Up to 4 months
  Proportion of respondents reporting a score of >3 on a two-item depression screening instrument (patient health questionnaire-2)
Medicine as a calling | Up to 4 months
  Composite measure comprised of 15 statements using true/false response scale to assess view of work as "calling," "career," or "job"
Medical learning environment that supports professionalism | Up to 4 months
  Composite measure comprised of 13 statements using 5-point Likert-type response scale (strongly disagree-strongly agree) to assess experiences of medical professionalism in medical students' learning environments

CONTACTS AND LOCATIONS:
Overall Officials: Audiey Kao, MD, PhD, Principal Investigator — American Medical Association

REFERENCES:
- [Background] Shearer DA. Management styles and motivation. Radiol Manage. 2012 Sep-Oct;34(5):47-52. PMID 23130386
- [Background] Wright SM, Beasley BW. Motivating factors for academic physicians within departments of medicine. Mayo Clin Proc. 2004 Sep;79(9):1145-50. doi: 10.4065/79.9.1145. PMID 15357036
- [Background] Williams GC, Rodin GC, Ryan RM, Grolnick WS, Deci EL. Autonomous regulation and long-term medication adherence in adult outpatients. Health Psychol. 1998 May;17(3):269-76. doi: 10.1037//0278-6133.17.3.269. PMID 9619477
- [Background] Williams GC, Deci EL. Internalization of biopsychosocial values by medical students: a test of self-determination theory. J Pers Soc Psychol. 1996 Apr;70(4):767-79. doi: 10.1037//0022-3514.70.4.767. PMID 8636897
- [Background] Williams GC, Wiener MW, Markakis KM, Reeve J, Deci EL. Medical students' motivation for internal medicine. J Gen Intern Med. 1994 Jun;9(6):327-33. doi: 10.1007/BF02599180. PMID 8077997
- [Background] Cerasoli CP, Nicklin JM, Ford MT. Intrinsic motivation and extrinsic incentives jointly predict performance: a 40-year meta-analysis. Psychol Bull. 2014 Jul;140(4):980-1008. doi: 10.1037/a0035661. Epub 2014 Feb 3. PMID 24491020
- [Background] Gonzalez MG, Swanson DP, Lynch M, Williams GC. Testing satisfaction of basic psychological needs as a mediator of the relationship between socioeconomic status and physical and mental health. J Health Psychol. 2016 Jun;21(6):972-82. doi: 10.1177/1359105314543962. Epub 2014 Aug 7. PMID 25104782
- [Background] Murayama K, Matsumoto M, Izuma K, Matsumoto K. Neural basis of the undermining effect of monetary reward on intrinsic motivation. Proc Natl Acad Sci U S A. 2010 Dec 7;107(49):20911-6. doi: 10.1073/pnas.1013305107. Epub 2010 Nov 15. PMID 21078974
- [Background] Wrzesniewski A, Schwartz B, Cong X, Kane M, Omar A, Kolditz T. Multiple types of motives don't multiply the motivation of West Point cadets. Proc Natl Acad Sci U S A. 2014 Jul 29;111(30):10990-5. doi: 10.1073/pnas.1405298111. Epub 2014 Jun 30. PMID 24982165